CLINICAL TRIAL: NCT03521635
Title: A Two- Stage Multicenter, Open-label, Randomized, Active Controlled Parallel Group Study Comparing the Efficacy and Safety of Pramipexole SR Versus Pramipexole IR Administered Orally Over an 18-week Treatment on Nocturnal Symptoms in L-Dopa+ Treated Patients With Advanced Parkinson's Disease (PD)
Brief Title: The SUSTAIN Study Compares the Effects of Sustained and Immediate-release Pramipexole on the noctUrnal Symptoms of paTients With Advanced ParkInsoN's Disease Who Also Take L-Dopa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0248-0686
Record Dates: First submitted 2018-04-11; First posted 2018-05-11 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pramipexole SR (Experimental)
  Interventions: Drug: Pramipexole SR
- Pramipexole IR (Active Comparator)
  Interventions: Drug: Pramipexole IR

INTERVENTIONS:
Drug: Pramipexole SR — Tablets
  Other Names: MIRAPEX®/SIFROL
  Arms: Pramipexole SR
Drug: Pramipexole IR — Tablets
  Other Names: MIRAPEX®/SIFROL
  Arms: Pramipexole IR

SUMMARY:
The main objective of the study is to explore firstly, then further evaluate and confirm the efficacy between Pramipexole Sustained Release (SR) versus Pramipexole Immediate Release (IR) on nocturnal symptoms (as measured by the change from baseline to the end of the maintenance period in Parkinson's Disease Sleep Scale 2nd version (PDSS-2) score) in L-dopa+ treated patients with advanced Parkinson's disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with advanced idiopathic Parkinson's disease (PD) confirmed by at least bradykinesia and one of the following signs: resting tremor, rigidity.
* Diagnosed as Parkinson's disease, with at least 2 years' PD history.
* Of age ≥ 30 years at time of diagnosis.
* Modified Hoehn and Yahr stage of 2 to 4 at on-time.
* They must have clinically relevant sleep disturbances (i.e. Parkinson's Disease Sleep Scale 2nd version (PDSS-2) total score ≥18 at baseline).
* They must feel uncomfortable at night because they were unable to turn around in bed or move due to immobility (i.e. the scoring of question 9 in PDSS-2 ≥ 2, that means frequency is at least 2 to 3 days during the past week).
* They must have early morning off (i.e. the frequency of "feeling like bodily movements are poor when you wake up?" is at least 2 to 3 days during the past week).
* Patient must have motor fluctuations (at least 2 cumulative hours of off-time every day during waking hours, documented on a patient diary completed for 2 consecutive days before randomization visit).
* Patients must be treated with Levodopa combined with a Dopa-Decarboxylase-inhibitor (L-Dopa+) (i.e. standard and/or controlled release Levodopa/DDC inhibitor), or with a combination of L-Dopa+ and entacapone, at an optimized dose according to investigator's judgment, this dose being stable for at least 4 weeks prior to randomization visit.
* Patients must not have been treated with sustained release dopaminergic drug (i.e. sustained release Levodopa/Dopa-Decarboxylase (DDC) inhibitor) after supper, or any anti-PD medication after 9pm within 4 weeks prior to randomization visit.
* Patients must not have been treated with dopamine agonists within 4 weeks prior to randomization visit. A concomitant treatment with one or more of the following drugs will be allowed (at a stable dose for at least 4 weeks prior to randomization visit and the investigator does not intend to change this treatment during the treatment phase):

  * Anti-parkinsonian anticholinergics;
  * Selegiline, rasagiline, or other Monoamine Oxydase (MAO)-B-Inhibitor;
  * Amantadine;
  * Entacapone (or other Catechol-O-Methyltransferase (COMT)-Inhibitor).
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

Exclusion criteria:

* Secondary parkinsonian syndromes due to drugs (e.g., metoclopramide, flunarizine), metabolic disorders (e.g., Wilson's disease), encephalitis or degenerative diseases (e.g., progressive supranuclear palsy).
* Dementia, as defined by a Mini-Mental State Exam score < 24 at screening visit.
* Any psychiatric disorder according to DSM-V Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria that could prevent compliance or completion of the study and/or put the patient at risk if he/she takes part in the study.
* History of psychosis, except history of drug induced hallucinations (provided the investigator considers that participation to the trial would not represent a significant risk for the patient).
* History of deep brain stimulation.
* History of nucleus lesioning.
* Clinically significant electrocardiogram (ECG) abnormalities at screening visit, according to investigator's judgement.
* Clinically significant hypotension (i.e. supine systolic blood pressure < 90 mmHg) and/or symptomatic orthostatic hypotension (i.e. clinical symptoms of orthostatic hypotension associated with a decline ≥ 20 mmHg in systolic blood pressure and a decline ≥ 10 mmHg in diastolic blood pressure, at 1 minute after standing compared with the previous supine systolic and diastolic blood pressure obtained after 5 minutes of quiet rest) at screening or randomization visit.
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned within 12 months after screening, e.g. hip replacement.
* Any other clinically significant disease, whether treated or not, that could put the patient at risk or could prevent compliance or completion of the study.
* Serious Sleep Apnea Hypopnea Syndrome (i.e. the scoring of question 15 in Parkinson's Disease Sleep Scale 2nd version (PDSS-2)≥ 3, that means frequency is at least 4 to 5 days during the past week )
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Serum levels of Aspartate Aminotransferase (AST)(SGOT), Alanine Aminotransferase (ALT)(SGPT), alkaline phosphatases or total bilirubin >2 ULN (on screening lab test).
* Patients with a creatinine clearance < 50 mL/min (estimated by the local lab / the investigator using the Modification of Diet in Renal Disease (MDRD, please refer to Appendix 10.1), and calculated on screening lab test).
* Any hypnotic medication within 4 weeks prior to the randomization visit (i.e. diazepam, clonazepam, estazolam, alprazolam, zolpidem, etc.).
* Any medication (including intra-muscular formulations) with central dopaminergic antagonist activity within 4 weeks prior to the randomization visit (i.e. typical neuroleptics, atypical antipsychotics, reserpine, methyldopa, centrally-active antiemetics, etc.).
* Any of the following drugs within 4 weeks prior to randomization visit: methylphenidate, cinnarizine, amphetamines.
* Flunarizine within 3 months prior to randomization visit.
* Known hypersensitivity to Pramipexole or its excipients.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Previous enrolment in this trial.
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s).
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant in the trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Hospital, Beijing
  - West China Hospital, Chengdu
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - 2nd Affiliated Hosp Zhejiang University College of Medical, Hangzhou
  - Brain Hospital Affiliated to Nanjing Med University, Nanjing
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Hospital of Chinese Medical University, Shenyang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 2-stage open-label, randomised, active controlled parallel group study compared the efficacy and safety of Pramipexole Sustained Release versus Immediate Release administered orally over an 18-week treatment on nocturnal symptoms in patients on Levodopa combined with a Dopa-Decarboxylase-inhibitor with advanced Parkinson's disease.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Pramipexole Sustained Release: Tablets of Pramipexole sustained release (SR) with unit strength of 0.375 milligram (mg) and 0.75 mg were administered orally once daily at 7-9 pm before bedtime to achieve daily dose of 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg for a treatment period of 18 weeks. The dose of Pramipexole SR was titrated to an optimised level, to achieve a maximum therapeutic effect without intolerable side effects.
- Pramipexole Immediate Release: Tablets of Pramipexole immediate release (IR) with unit strength of 0.25 milligram (mg) and 1.0 mg were administered in equally divided doses three times per day to achieve a total daily dose of 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, the third dose at 7-9 pm before bedtime for a treatment period of 18 weeks.
  The dose of Pramipexole IR was titrated to an optimised level, to achieve a maximum therapeutic effect without intolerable side effects.
Period: Overall Study
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Started | 49 | 49
Completed | 45 | 43
Not Completed | 4 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Refused to complete study visit | 1 | 0
Not completed — Refused to continue trial medication | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Meet exclusion criteria | 0 | 1
Not completed — Patient not taken study medicine | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) was defined as all patients who were dispensed study medication and were documented to have at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (10.80) | 60.9 (8.83) | 61.0 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 28 | 31 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 49 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 49 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Parkinson's disease Sleep Scale 2nd version (PDSS-2) total score [Mean (Standard Deviation); unit: Score on scale] — Parkinson's disease Sleep Scale 2nd version (PDSS-2) consists of 15 questions about various sleep and nocturnal disturbances which are to be rated by the patients using one of five categories, from 0 (never) to 4 (very often).
  Patients were asked to rate the severity of each question based on their experience during the past week (7 days) from 0 (Never) to 4 (Very often, that meant 6 to 7 days a week). PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance).
  Score on scale | 27.8 (6.45) | 29.2 (8.53) | 28.5 (7.56)
Parkinson's disease Questionnaire (PDQ) -8 score [Mean (Standard Deviation); unit: Score on a scale] — The PDQ-8 is a self-reported questionnaire consisting of 8 questions regarding the subject's disease symptoms, each item ranging from 0 to 4, and the responses consist of 0=Never, 1=Occasionally, 2=Sometimes, 3=Often, and 4=Always or cannot do at all, total score ranging from 0 (never have problems/issues) to 32 (always have problems or cannot do at all).
  Score on a scale | 11.3 (4.83) | 10.5 (4.99) | 10.9 (4.90)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 18 in Parkinson's Disease Sleep Scale 2nd Version (PDSS-2) Total Score
Description: Parkinson's disease Sleep Scale 2nd version (PDSS-2) consists of 15 questions about various sleep and nocturnal disturbances which are to be rated by the patients using one of five categories, from 0 (never) to 4 (very often). Patients were asked to rate the severity of each question based on their experience during the past week (7 days) from 0 (Never) to 4 (Very often, that meant 6 to 7 days a week). PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance).
Time Frame: Baseline and Week 18
Population: Full analysis set (FAS) was defined as all patients who were randomised to treatment and received at least one dose of study drug and providing a baseline and at least one PDSS-2 total score measurement in maintenance period.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Score on a scale | -13.7 (1.16) | -14.4 (1.20)
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of PDSS-2 score were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.688, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = 0.7, 95% CI 2-sided [-2.7 to 4.0], Standard Error of Mean 1.68 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release

2. Secondary Outcome: Nocturnal Hypokinesia Questionnaire (NHQ) Score (Change From Baseline)
Description: The Nocturnal Hypokinesia Questionnaire (NHQ) is designed to assess hypokinesia symptoms in night in Parkinson's disease (PD) patients, composed of two sections. Section 1 is assessed by PD patients with 10 one-point items evaluating "turning over in bed", "getting out of bed", "parkinsonian motor symptoms", and "others". Section 2 is assessed by spouses or caregivers who are with the patients during the night with 10 one-point items evaluating the same aspects as Section 1. The score for each section is by summing up points from the items in the respective section. Score of each of the two Sections is from 0 to 10, with a higher score indicating worse symptoms. The score was reported by section: Section 1 by patients, Section 2 by caregivers.
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Score on a scale
  By patients (Section 1) | -1.9 (0.35) | -1.7 (0.36)
  By caregivers (Section 2): number analyzed (Participants) | 13 | 11
  By caregivers (Section 2) | -1.4 (0.61) | -0.6 (0.67)
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of NHQ score by patients were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.690, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.2, 95% CI 2-sided [-1.2 to 0.8], Standard Error of Mean 0.51 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release
Statistical Analysis 2: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of NHQ score by caregivers were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.376, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.8, 95% CI 2-sided [-2.7 to 1.1], Standard Error of Mean 0.91 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release

3. Secondary Outcome: Scale for Outcomes in Parkinson's Disease (SCOPA)-Sleep Score (Change From Baseline)
Description: SCOPA-Sleep score is composed of three parts: a night-time scale (5 item scale with 4 Response Options (0-not at all to 3-very much) addressing night time disturbances. Total night-time scale score runs from 0 to 15, with a higher score indicating more severe problems, a single-item about perceived quality of nocturnal sleep (7-point scale ranging from slept very well to slept very badly.), and a daytime sleepiness scale (6 items with 4 Response options, from 0 (never) to 3 (often), and a maximum total score of 18.).
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Score on a scale
  Night-time sleep score | -3.8 (0.46) | -3.2 (0.47)
  Overall night sleep score | -1.9 (0.20) | -1.6 (0.21)
  Daytime sleepiness score | -1.4 (0.34) | -0.9 (0.35)
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of SCOPA-Sleep night-time sleep score were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.333, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.6, 95% CI 2-sided [-1.9 to 0.7], Standard Error of Mean 0.66 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release
Statistical Analysis 2: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of SCOPA-Sleep overall night sleep score were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.374, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.3, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.29 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release
Statistical Analysis 3: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of SCOPA-Sleep daytime sleepiness score were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.352, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.5, 95% CI 2-sided [-1.4 to 0.5], Standard Error of Mean 0.49 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release

4. Secondary Outcome: Early Morning Off (EMO) Score (Change From Baseline)
Description: The EMO is measured by the question of "do you feel like your bodily movements are poor when you wake up?" Patients answered this question according to the frequency during the previous one week by scoring from 0 ("never") to 4 ("very often" or "6 to 7 days a week").
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Score on a scale | -1.8 (0.18) | -1.5 (0.18)
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of EMO sore were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.259, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.3, 95% CI 2-sided [-0.8 to 0.2], Standard Error of Mean 0.26 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release

5. Secondary Outcome: Responder Rate for Parkinson's Disease Sleep Scale 2nd Version (PDSS-2) Total Score<18
Description: Parkinson's disease Sleep Scale 2nd version (PDSS-2) consists of 15 questions about various sleep and nocturnal disturbances which are to be rated by the patients using one of five categories, from 0 (never) to 4 (very often) based on their experience during the past week. PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance). The PDSS-2 total score less < 18 were compared between groups.
Time Frame: At Week 18
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Percentage of participants | 73.3 [58.1 to 85.4] | 72.1 [56.3 to 84.7]
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Logistic regression analyses for responder rate at week 18 of PDSS-2 score <18 were performed with treatment and baseline as the independent variables; Test type: Other; p = 0.9373, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.36 to 2.54] — The odds ratio (OR) between Pramipexole Sustained Release and Pramipexole Immediate Release groups

6. Secondary Outcome: Responder Rate for Early Morning Off (EMO) Score
Description: The responder of EMO is the patient with an improvement of at least 1 comparing to his/her baseline condition. The EMO is measured by the question of "do you feel like your bodily movements are poor when you wake up?" Patients answered this question according to the frequency during the previous one week by scoring from 0 ("never") to 4 ("very often" or "6 to 7 days a week").
Time Frame: At Week 18
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Percentage of participants | 86.7 [73.2 to 94.9] | 76.7 [61.4 to 88.2]
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Logistic regression analyses for responder rate at week 18 of EMO score were performed with treatment and baseline as the independent variables; Test type: Other; p = 0.1611, Regression, Logistic; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.73 to 7.49] — The odds ratio (OR) between Pramipexole Sustained Release and Pramipexole Immediate Release groups

7. Secondary Outcome: The Parkinson's Disease Questionnaire (PDQ)-8 Score (Change From Baseline)
Description: The PDQ-8 is a self-reported questionnaire consisting of 8 questions regarding the subject's disease symptoms. The total score summed up the items together and transformed onto a score from 0 (never have problems/issues) to 100 (always have problems or cannot do at all).
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Score on a scale | -4.1 (0.60) | -3.5 (0.62)
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of PDQ-8 score were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.517, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = -0.6, 95% CI 2-sided [-2.3 to 1.2], Standard Error of Mean 0.87 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release

8. Secondary Outcome: Responder Rate for Clinical Global Impression of Improvement (CGI-I)
Description: The responder of CGI-I is the patient rated of any improvement (1 = Very much better, 2 = Much better, or 3 = A little better). The CGI-I was rated (from 1: very much improved, to 7: very much worse) by the same evaluator to assess the overall status of Parkinson's disease.
Time Frame: At Week 18
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Percentage of participants | 95.6 [84.9 to 99.5] | 86.0 [72.1 to 94.7]
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Logistic regression analyses for responder rate at week 18 of CGI-I were performed with treatment as the independent variable; Test type: Other; p = 0.2374, Regression, Logistic; Odds Ratio (OR) = 3.44, 95% CI 2-sided [0.57 to 36.85] — The odds ratio (OR) between Pramipexole Sustained Release and Pramipexole Immediate Release groups

9. Secondary Outcome: Responder Rate for Patient Global Impression of Improvement (PGI-I)
Description: The responder of PGI-I is the patient rated of any improvement (1 = Very much better, 2 = Much better, or 3 = A little better). The PGI-I scale is a patient-rated instrument (from 1: very much better, to 7: very much worse) which was used to measure the improvement of the patient's Parkinson disease symptoms throughout the study.
Time Frame: At Week 18
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Percentage of participants | 95.6 [84.9 to 99.5] | 86.0 [72.1 to 94.7]
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Logistic regression analyses for responder rate at week 18 of PGI-I were performed with treatment as the independent variable; Test type: Other; p = 0.2374, Regression, Logistic; Odds Ratio (OR) = 3.44, 95% CI 2-sided [0.57 to 36.85] — The odds ratio (OR) between Pramipexole Sustained Release and Pramipexole Immediate Release groups

10. Secondary Outcome: Epworth Sleepiness Scale (ESS) Score (Change From Baseline)
Description: The ESS is a patient-rated scale about how likely one is to fall asleep during situations of passive and inconsequential to active. The total score ranges from 0-24 where higher values indicate greater daytime sleepiness.
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
Number analyzed (Participants) | 45 | 43
Score on a scale | -2.4 (0.54) | -2.6 (0.56)
Statistical Analysis 1: Comparison: Pramipexole Sustained Release vs Pramipexole Immediate Release; Mean changes from baseline of ESS score were analysed using a restricted maximum likelihood (REML) - based repeated measures approach. Analyses included the fixed, categorical effects of treatment, visit in the maintenance period, and treatment-by-visit interaction, and the continuous, fixed covariates of baseline and baseline-by-visit interaction; Test type: Other; p = 0.820, REML-based repeated measures approach; Restricted maximum likelihood (REML) - based repeated measures approach was applied; Adjusted mean difference = 0.2, 95% CI 2-sided [-1.4 to 1.7], Standard Error of Mean 0.79 — Mean difference was calculated as Pramipexole Sustained Release minus Pramipexole immediate Release

ADVERSE EVENTS:
Time Frame: From randomisation through end of treatment until end of follow up visit, up to 18 weeks + 2 days.
Description: Treated set (TS) was defined as all patients who were dispensed study medication and were documented to have at least one dose of investigational treatment.
Arm/Group | Pramipexole Sustained Release | Pramipexole Immediate Release
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/49
Other Adverse Events (participants affected / at risk) | 4/49 | 7/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Sustained Release (N=49) | Pramipexole Immediate Release (N=49)
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Sustained Release (N=49) | Pramipexole Immediate Release (N=49)
Dizziness (Nervous system disorders) | 3 | 3
Dyskinesia (Nervous system disorders) | 1 | 3
Somnolence (Nervous system disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
According to the study results, the decision was made to stop transitioning to Stage II. Therefore, only results of Stage I were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03521635/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT03521635/SAP_001.pdf